CLINICAL TRIAL: NCT00637377
Title: A Randomized, Double Masked, Active Controlled, Phase 3 Study of the Efficacy, Safety, and Tolerability of Repeated Doses of Intravitreal VEGF Trap in Subjects With Neovascular Age-related Macular Degeneration (AMD)
Brief Title: Vascular Endothelial Growth Factor (VEGF) Trap-Eye: Investigation of Efficacy and Safety in Wet Age-Related Macular Degeneration (AMD)
Acronym: VIEW 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 91689; 2007-000583-25 (EudraCT Number)
Record Dates: First submitted 2008-03-12; First posted 2008-03-18 (Estimated); Results first posted 2012-01-23 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-11

CONDITIONS: Macular Degeneration
Keywords: Eye diseases; Vision Impairment and Blindness; Eyes and Vision; Seniors; Neovascular Age-Related Macular Degeneration (AMD); Retinal Disease
MeSH Terms: conditions — Macular Degeneration; Eye Diseases; Vision Disorders; Blindness; Retinal Diseases | interventions — Ranibizumab; aflibercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Ranibizumab 0.5mg Q4 (Active Comparator): Participants received a 0.5 mg dose of Ranibizumab via intravitreal (IVT) injection administered every 4 weeks for the first year. Thereafter a dose may be administered as frequently as every 4 weeks, but no less frequently than every 12 weeks.
  Interventions: Drug: Ranibizumab
- Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg Q4 (Experimental): Participants received a 2.0 mg dose of Aflibercept Injection administered every 4 weeks for the first year. Thereafter a dose may be administered as frequently as every 4 weeks, but no less frequently than every 12 weeks.
  Interventions: Biological: Aflibercept Injection (EYLEA, VEGF Trap-Eye, BAY86-5321)
- Aflibercept Injection (EYLEA, VEGF Trap-Eye) 0.5mg Q4 (Experimental): Participants received a 0.5 mg dose of Aflibercept Injection administered every 4 weeks for the first year. Thereafter a dose may be administered as frequently as every 4 weeks, but no less frequently than every 12 weeks.
  Interventions: Biological: Aflibercept Injection (EYLEA, VEGF Trap-Eye, BAY86-5321)
- Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg Q8 (Experimental): Participants received a 2.0 mg dose of Aflibercept Injection administered every 8 weeks (including one additional 2,0 mg dose at Week 4) for the first year. Thereafter a dose may be administered as frequently as every 4 weeks, but no less frequently than every 12 weeks.
  Interventions: Biological: Aflibercept Injection (EYLEA, VEGF Trap-Eye, BAY86-5321)

INTERVENTIONS:
Drug: Ranibizumab — Participants received a 0.5 mg dose of Ranibizumab via intravitreal (IVT) injection administered every 4 weeks for the first year. Thereafter a dose may be administered as frequently as every 4 weeks, but no less frequently than every 12 weeks.
  Arms: Ranibizumab 0.5mg Q4
Biological: Aflibercept Injection (EYLEA, VEGF Trap-Eye, BAY86-5321) — Participants received a 2.0 mg dose of Aflibercept Injection administered every 4 weeks for the first year. Thereafter a dose may be administered as frequently as every 4 weeks, but no less frequently than every 12 weeks.
  Arms: Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg Q4
Biological: Aflibercept Injection (EYLEA, VEGF Trap-Eye, BAY86-5321) — Participants received a 0.5 mg dose of Aflibercept Injection administered every 4 weeks for the first year. Thereafter a dose may be administered as frequently as every 4 weeks, but no less frequently than every 12 weeks.
  Arms: Aflibercept Injection (EYLEA, VEGF Trap-Eye) 0.5mg Q4
Biological: Aflibercept Injection (EYLEA, VEGF Trap-Eye, BAY86-5321) — Participants received a 2.0 mg dose of Aflibercept Injection administered every 8 weeks (including one additional 2,0 mg dose at Week 4) for the first year. Thereafter a dose may be administered as frequently as every 4 weeks, but no less frequently than every 12 weeks.
  Arms: Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg Q8

SUMMARY:
This study is a phase III, double-masked, randomized, study of the efficacy and safety of VEGF Trap-Eye in patients with neovascular age-related macular degeneration. Approximately 1200 patients will be randomized in Europe, Asia, Japan, Australia and South America.

DETAILED DESCRIPTION:
Data of this trial ("VIEW 2") was pooled with data of a sister trial ("VIEW 1", NCT00509795), and an integrated analyses of the combined data was performed.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Men and women >/=50 years of age.
* Active primary or recurrent subfoveal CNV lesions secondary to AMD, including juxtafoveal lesions that affect the fovea as evidenced by Fluorescein angiography (FA) in the study eye.
* ETDRS Best-Corrected Visual Acuity letter score of 73 to 25 (= Acuity of 20/40 to 20/320) in the study eye at 4 meters.
* Willing, committed, and able to return for ALL clinic visits and complete all study-related procedures.
* Able to read, (or, if unable to read due to visual impairment, be read to verbatim by the person administering the informed consent or a family member) understand and willing to sign the informed consent form.

Exclusion Criteria:

* Any prior ocular (in the study eye) or systemic treatment or surgery for neovascular AMD, except dietary supplements or vitamins.
* Any prior or concomitant therapy with another investigational agent to treat neovascular AMD in the study eye.
* Any prior treatment with anti-VEGF agents in the study eye.
* Total lesion size >12 disc areas (30.5 mm, including blood, scars and neovascularization) as assessed by FA in the study eye.
* Subretinal hemorrhages that is either 50% or more of the total lesion area, or if the blood is under the fovea and is 1 or more disc areas in size in the study eye (if the blood is under the fovea, then the fovea must be surrounded by 270 degrees by visible CNV).
* Scar or fibrosis making up >50% of the total lesion in the study eye.
* Scar, fibrosis, or atrophy involving the center of the fovea in the study eye.
* Presence of retinal pigment epithelial tears or rips involving the macula in the study eye.
* History of any vitreous hemorrhage within 4 weeks prior to Visit 1 in the study eye.
* Presence of other causes of CNV in the study eye.
* Prior vitrectomy in the study eye.
* History of retinal detachment or treatment or surgery for retinal detachment in the study eye.
* Any history of macular hole of stage 2 and above in the study eye.
* Any intraocular or periocular surgery within 3 months of Day 1 on the study eye, except lid surgery, which may not have taken place within 1 month of Day 1, as long as it is unlikely to interfere with the injection.
* History or clinical evidence of diabetic retinopathy, diabetic macular edema or any retinal vascular disease other than AMD in either eye.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1240 (Actual)
Dates: Start 2008-04; Primary Completion 2010-09 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (158):
- Argentina (3):
  - Buenos Aires, Ciudad Auton. de Buenos Aires
  - Córdoba, Córdoba Province
  - Rosario, Santa Fe Province
- Australia (7):
  - Chatswood, New South Wales
  - Sydney, New South Wales
  - Westmead, New South Wales
  - East Melbourne, Victoria
  - Parkville, Victoria
  - Nedlands, Western Australia
  - Parramatta
- Austria (3):
  - Innsbruck
  - Linz
  - Vienna
- Liège, Belgium
- Brazil (3):
  - Ribeirão Preto, São Paulo
  - São Paulo, São Paulo
  - Minas Gerais
- Colombia (3):
  - Medellín, Antioquia
  - Bogotá, Bogota D.C.
  - Cali, Cauca Department
- Czechia (4):
  - Brno
  - Olomouc
  - Prague
  - Ústí nad Labem
- France (8):
  - Paris, Cedex 12
  - Nantes, Cedex 1
  - Besançon
  - Bordeaux
  - Dijon
  - Lyon
  - Marseille
  - Paris
- Germany (20):
  - Freiburg im Breisgau, Baden-Wurttemberg
  - Heidelberg, Baden-Wurttemberg
  - Tübingen, Baden-Wurttemberg
  - München, Bavaria
  - Regensburg, Bavaria
  - Hamburg, Hamburg
  - Darmstadt, Hesse
  - Aachen, North Rhine-Westphalia
  - Bonn, North Rhine-Westphalia
  - Cologne, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
  - Münster, North Rhine-Westphalia
  - Ludwigshafen am Rhein, Rhineland-Palatinate
  - Mainz, Rhineland-Palatinate
  - Homburg, Saarland
  - Dresden, Saxony
  - Leipzig, Saxony
  - Kiel, Schleswig-Holstein
  - Lübeck, Schleswig-Holstein
  - Berlin, State of Berlin
- Hungary (2):
  - Budapest
  - Veszprém
- India (14):
  - Ahemedabad - 4, Gujarat
  - Wadala, Mumbai, Maharashtra
  - Chennai, Tamil Nadu
  - Coimbatore, Tamil Nadu
  - Madurai, Tamil Nadu
  - Pondicherry, Tamil Nadu
  - Bangalore
  - Chandigarh
  - Hyderabad
  - Kerala
  - Kolkata
  - Mumbai
  - New Delhi
  - Orissa
- Israel (10):
  - Haifa, Israel
  - Kfar Saba, Israel
  - Petah Tikva, Israel
  - Zrifin, Israel
  - Afula
  - Beersheba
  - Jerusalem
  - Rehovot
  - Tel Aviv
  - Tel Litwinsky
- Italy (11):
  - Ancona
  - Bari
  - Catania
  - Genova
  - Milan
  - Padua
  - Roma
  - Torino
  - Udine
  - Varese
  - Verona
- Japan (14):
  - Nagoya, Aichi-ken
  - Urayasu, Chiba
  - Fukuoka, Fukuoka
  - Fukushima, Fukushima
  - Maebashi, Gunma
  - Sapporo, Hokkaido
  - Kita, Kagawa-ken
  - Kagoshima, Kagoshima-ken
  - Kyoto, Kyoto
  - Hirakata, Osaka
  - Suita, Osaka
  - Ōtsu, Shiga
  - Chiyoda-ku, Tokyo
  - Shinjuku-ku, Tokyo
- Riga, Latvia
- Mexico (7):
  - Chihuahua City, Chihuahua
  - Zapopan, Jalisco
  - Mexico City, Mexico City
  - Monterrey, Nuevo León
  - Metepec, State of Mexico
  - Mexico City
  - México D.F.
- Netherlands (5):
  - Leiden, ZA
  - Amsterdam
  - Groningen
  - Nijmegen
  - Rotterdam
- Poland (7):
  - Bydgoszcz
  - Gdansk
  - Katowice
  - Poznan
  - Warsaw
  - Warszaa
  - Wroclaw
- Portugal (2):
  - Coimbra
  - Porto
- Singapore, Singapore
- Slovakia (2):
  - Banská Bystrica
  - Bratislava
- South Korea (3):
  - Seongnam, Gyeonggido
  - Incheon
  - Seoul
- Spain (11):
  - Santiago de Compostela, A Coruña
  - Alicante, Alicante
  - Madrid, Madrid
  - Pamplona, Navarre
  - Oviedo, Principality of Asturias
  - Barcelona
  - Madrid
  - Málaga
  - Seville
  - Valencia
  - Valladolid
- Sweden (3):
  - Linköping
  - Örebro
  - Stockholm
- Switzerland (4):
  - Basel
  - Bern
  - Geneva
  - Zurich
- United Kingdom (9):
  - Southampton, Hampshire
  - Camberley, Surrey
  - Aberdeen
  - Belfast
  - Birmingham
  - Liverpool
  - London
  - Plymouth
  - Torquay

REFERENCES:
- [Result] Heier JS, Brown DM, Chong V, Korobelnik JF, Kaiser PK, Nguyen QD, Kirchhof B, Ho A, Ogura Y, Yancopoulos GD, Stahl N, Vitti R, Berliner AJ, Soo Y, Anderesi M, Groetzbach G, Sommerauer B, Sandbrink R, Simader C, Schmidt-Erfurth U; VIEW 1 and VIEW 2 Study Groups. Intravitreal aflibercept (VEGF trap-eye) in wet age-related macular degeneration. Ophthalmology. 2012 Dec;119(12):2537-48. doi: 10.1016/j.ophtha.2012.09.006. Epub 2012 Oct 17. PMID 23084240
- [Result] Schmidt-Erfurth U, Kaiser PK, Korobelnik JF, Brown DM, Chong V, Nguyen QD, Ho AC, Ogura Y, Simader C, Jaffe GJ, Slakter JS, Yancopoulos GD, Stahl N, Vitti R, Berliner AJ, Soo Y, Anderesi M, Sowade O, Zeitz O, Norenberg C, Sandbrink R, Heier JS. Intravitreal aflibercept injection for neovascular age-related macular degeneration: ninety-six-week results of the VIEW studies. Ophthalmology. 2014 Jan;121(1):193-201. doi: 10.1016/j.ophtha.2013.08.011. Epub 2013 Sep 29. PMID 24084500
- [Derived] Lukacs R, Schneider M, Nagy ZZ, Sandor GL, Kaan K, Asztalos A, Enyedi L, Pek G, Barcsay G, Szabo A, Borbandy A, Kovacs I, Resch MD, Papp A. Seven-year outcomes following intensive anti-vascular endothelial growth factor therapy in patients with exudative age-related macular degeneration. BMC Ophthalmol. 2023 Mar 17;23(1):110. doi: 10.1186/s12886-023-02843-2. PMID 36932356
- [Derived] Moshfeghi DM, Thompson D, Saroj N. Changes in neovascular activity following fixed dosing with an anti-vascular endothelial growth factor agent over 52 weeks in the phase III VIEW 1 and VIEW 2 studies. Br J Ophthalmol. 2020 Sep;104(9):1223-1227. doi: 10.1136/bjophthalmol-2019-315021. Epub 2019 Dec 11. PMID 31826853
- [Derived] Yuzawa M, Fujita K, Wittrup-Jensen KU, Norenberg C, Zeitz O, Adachi K, Wang EC, Heier J, Kaiser P, Chong V, Korobelnik JF. Improvement in vision-related function with intravitreal aflibercept: data from phase 3 studies in wet age-related macular degeneration. Ophthalmology. 2015 Mar;122(3):571-8. doi: 10.1016/j.ophtha.2014.09.024. Epub 2014 Nov 6. PMID 25439429
- [Derived] Ogura Y, Terasaki H, Gomi F, Yuzawa M, Iida T, Honda M, Nishijo K, Sowade O, Komori T, Schmidt-Erfurth U, Simader C, Chong V; VIEW 2 Investigators. Efficacy and safety of intravitreal aflibercept injection in wet age-related macular degeneration: outcomes in the Japanese subgroup of the VIEW 2 study. Br J Ophthalmol. 2015 Jan;99(1):92-7. doi: 10.1136/bjophthalmol-2014-305076. Epub 2014 Aug 8. PMID 25107900
- See also: Click here to view the data of the twin trial conducted by the collaboration partner. — http://clinicaltrials.gov/ct2/show/NCT00509795?term=NCT00509795;rank=1
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 186 study centers in 26 countries. Recruitment period: 21 Apr 2008 - 4 Sep 2009.
Pre-assignment Details: 2031 participants were screened, 1240 were randomized and 1204 received at least 1 dose of study drug. 1204 participants were included in the Safety-Analysis Set (SAS). 1202 participants with at least 1 post-baseline measurement were included in the Full-Analysis Set (FAS).
Groups:
- Ranibizumab 0.5mg Q4: Participants received a dose of 0.5 mg Ranibizumab every 4 weeks for the first year (intravitreal [IVT] injection). Thereafter a dose may be administered as frequently as every 4 weeks, but no less frequently than every 12 weeks.
- Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg Q4: Participants received a dose of 2.0 mg Aflibercept Injection every 4 weeks for the first year (intravitreal [IVT] injection). Thereafter a dose may be administered as frequently as every 4 weeks, but no less frequently than every 12 weeks.
- Aflibercept Injection (EYLEA, VEGF Trap-Eye) 0.5mg Q4: Participants received a dose of 0.5 mg Aflibercept Injection every 4 weeks for the first year (intravitreal [IVT] injection). Thereafter a dose may be administered as frequently as every 4 weeks, but no less frequently than every 12 weeks.
- Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg Q8: Participants received a dose of 2.0 mg Aflibercept Injection every 8 weeks (including one additional 2.0 mg dose at Week 4) for the first year (IVT injection) and were to receive sham injections at interim monthly visits. During the second year, participants received 2.0 mg aflibercept as frequently as every 4 weeks, but no less frequently than every 12 weeks.
Period: Overall Study
Arm/Group | Ranibizumab 0.5mg Q4 | Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg Q4 | Aflibercept Injection (EYLEA, VEGF Trap-Eye) 0.5mg Q4 | Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg Q8
Started | 303 | 313 | 311 | 313
Participants Received Treatment | 291 (safety population) | 309 (safety population) | 297 (safety population) | 307 (safety population)
Participants Treated (FAS) | 291 | 309 | 296 | 306
Completed | 276 | 281 | 274 | 284
Not Completed | 27 | 32 | 37 | 29
Not completed — Adverse Event | 2 | 6 | 8 | 9
Not completed — Death | 1 | 3 | 2 | 1
Not completed — Lack of Efficacy | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 4 | 1 | 2 | 2
Not completed — Protocol Violation | 2 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 11 | 15 | 13 | 11
Not completed — Other (no further information available) | 7 | 6 | 10 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranibizumab 0.5mg Q4 | Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg Q4 | Aflibercept Injection (EYLEA, VEGF Trap-Eye) 0.5mg Q4 | Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg Q8 | Total
Number analyzed (Participants) | 291 | 309 | 296 | 306 | 1202
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.0 (9.0) | 74.1 (8.5) | 74.7 (8.6) | 73.8 (8.6) | 73.9 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Information retrieved from all baseline participants.
  Participants
    Female | 169 | 176 | 147 | 175 | 667
    Male | 122 | 133 | 149 | 131 | 535
Ethnicity [Number; unit: participants] — Information retrieved from all baseline participants.
  participants
    Not Hispanic or Latino | 239 | 259 | 241 | 251 | 990
    Hispanic or Latino | 52 | 50 | 55 | 55 | 212
Race [Number; unit: participants] — Information retrieved from all baseline participants.
  participants
    White | 213 | 226 | 219 | 217 | 875
    Black or African American | 1 | 0 | 1 | 2 | 4
    Asian | 60 | 67 | 61 | 69 | 257
    Missing | 17 | 16 | 15 | 18 | 66
National Eye Institute 25-item Visual Function Questionnaire (NEI VFQ-25) total score [Mean (Standard Deviation); unit: scores on a scale] — Information retrieved from 1201/1202 baseline participants. The possible range of the NEI VFQ-25 total score is between 0 (worst possible) and 100 (best possible).
  scores on a scale | 72.90 (19.09) | 70.27 (19.41) | 74.04 (18.22) | 71.30 (19.06) | 72.10 (18.99)
Area of Choroidal Neovascularization (CNV) [Mean (Standard Deviation); unit: mm^2] — Information retrieved from 1200/1202 baseline participants.
  mm^2 | 7.59 (5.34) | 8.25 (5.77) | 7.70 (5.26) | 7.75 (5.52) | 7.83 (5.48)
Baseline lesion type [Number; unit: participants] — Information retrieved from 1197/1202 baseline participants.
  participants
    Predominantly classic | 70 | 72 | 80 | 88 | 310
    Minimally classic | 104 | 112 | 103 | 106 | 425
    Occult | 116 | 123 | 113 | 110 | 462
    Missing | 1 | 2 | 0 | 2 | 5
Baseline total lesion size [Mean (Standard Deviation); unit: mm^2] — Information retrieved from 1198/1202 baseline participants.
  mm^2 | 8.01 (5.74) | 8.72 (6.14) | 8.17 (5.51) | 8.22 (5.87) | 8.28 (5.82)
Best Corrected Visual Acuity (BCVA), assessed by ETDRS chart [Mean (Standard Deviation); unit: Letters correctly read] — Information retrieved from all baseline participants. Only participants with a ETDRS (Early Treatment Diabetic Retinopathy Study) Best Corrected Visual Acuity letter score of 73 to 25 (= Acuity of 20/40 to 20/320) in the study eye at 4 meters were included; a higher score represents better functioning.
  Letters correctly read | 53.8 (13.5) | 52.8 (13.9) | 51.6 (14.2) | 51.6 (13.9) | 52.4 (13.9)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Maintained Vision at Week 52 - Last Observation Carried Forward (LOCF)
Description: Maintenance of vision was defined as a loss of < 15 letters in the ETDRS (Early Treatment Diabetic Retinopathy Study) letter score (defined study baseline range of ETDRS Best Corrected Visual Acuity letter score of 73 to 25 (= Acuity of 20/40 to 20/320) in the study eye; a higher score represents better functioning.
  Nominator = (Number of participants who maintained vision * 100); Denominator = Number of participants analyzed.
Time Frame: At week 52
Population: Per-Protocol Set (PPS); imputation technique: LOCF
Measure: Number; unit: Percentage of participants
Arm/Group | Ranibizumab 0.5mg Q4 | Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg Q4 | Aflibercept Injection (EYLEA, VEGF Trap-Eye) 0.5mg Q4 | Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg Q8
Number analyzed (Participants) | 269 | 274 | 268 | 270
Percentage of participants | 94.42 | 95.62 | 96.27 | 95.56
Statistical Analysis 1: Comparison: Ranibizumab 0.5mg Q4 vs Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg Q4; null hypothesis: pi ≤ pc-delta where pi is the probability that a participant maintained vision at week 52 under Aflibercept 2mg Q4, pc is the probability that a participant maintained vision at week 52 under Ranibizumab 0.5mg Q4 and delta is the non-inferiority margin. The null hypothesis is tested calculating a two-sided 95 % confidence using normal approximation of the difference of percentages of participants maintaining vision at week 52 (Ranibizumab 0.5mg Q4 minus Aflibercept 2mg Q4); Test type: Non-Inferiority or Equivalence — The non-inferiority margin is set to 10. The power is 90 % according to the sample size estimation of the study protocol; Risk Difference (RD) = -1.20, 95% CI 2-sided [-4.86 to 2.46] — The difference is calculated as Ranibizumab minus Aflibercept. A negative value favors the Aflibercept 2mg Q4 group. As adjustment of multiple comparisons a conditional sequence of statistical hypotheses is used with alpha = 0.05
Statistical Analysis 2: Comparison: Ranibizumab 0.5mg Q4 vs Aflibercept Injection (EYLEA, VEGF Trap-Eye) 0.5mg Q4; null hypothesis: pi ≤ pc-delta where pi is the probability that a participant maintained vision at week 52 under Aflibercept 0.5mg Q4, pc is the probability that a participant maintained vision at week 52 under Ranibizumab 0.5mg Q4 and delta is the non-inferiority margin. The null hypothesis is tested calculating a two-sided 95 % confidence using normal approximation of the difference of percentages of participants maintaining vision at week 52 (Ranibizumab 0.5mg Q4 minus Aflibercept 0.5mg Q4); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Risk Difference (RD) = -1.84, 95% CI 2-sided [-5.40 to 1.71] — The difference is calculated as Ranibizumab minus Aflibercept. A negative value favors the Aflibercept 0.5mg Q4 group. As adjustment of multiple comparisons a conditional sequence of statistical hypotheses is used with alpha = 0.05
Statistical Analysis 3: Comparison: Ranibizumab 0.5mg Q4 vs Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg Q8; null hypothesis: pi ≤ pc-delta where pi is the probability that a participant maintained vision at week 52 under Aflibercept 2mg Q8, pc is the probability that a participant maintained vision at week 52 under Ranibizumab 0.5mg Q4 and delta is the non-inferiority margin. The null hypothesis is tested calculating a two-sided 95 % confidence using normal approximation of the difference of percentages of participants maintaining vision at week 52 (Ranibizumab 0.5mg Q4 minus Aflibercept 2mg Q8); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Risk Difference (RD) = -1.13, 95% CI 2-sided [-4.81 to 2.55] — The difference is calculated as Ranibizumab minus Aflibercept. A negative value favors the Aflibercept 2mg Q8 group. As adjustment of multiple comparisons a conditional sequence of statistical hypotheses is used with alpha = 0.05

2. Secondary Outcome: Mean Change From Baseline in Best Corrected Visual Acuity (BCVA) as Measured by ETDRS Letter Score at Week 52 - LOCF
Description: Defined study baseline range of ETDRS Best Corrected Visual Acuity letter score of 73 to 25 (= Acuity of 20/40 to 20/320) in the study eye; a higher score represents better functioning.
Time Frame: Baseline and at week 52
Population: Full-Analysis Set (FAS); imputation technique: LOCF
Measure: Mean (Standard Deviation); unit: Letters correctly read
Arm/Group | Ranibizumab 0.5mg Q4 | Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg Q4 | Aflibercept Injection (EYLEA, VEGF Trap-Eye) 0.5mg Q4 | Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg Q8
Number analyzed (Participants) | 291 | 309 | 296 | 306
Letters correctly read | 9.4 (13.5) | 7.6 (12.6) | 9.7 (14.1) | 8.9 (14.4)
Statistical Analysis 1: Comparison: Ranibizumab 0.5mg Q4 vs Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg Q4; The pairwise comparison is performed as contrast statement in the analysis of covariance model with treatment group as fixed factor (all 4 treatment groups) and the baseline ETDRS letter score as covariate. The null hypothesis is that both mean changes are equal; Test type: Superiority or Other; p = 0.076, ANCOVA — as adjustment of multiple comparisons a conditional sequence of statistical hypotheses (a-priori ordered hypotheses) is used with alpha = 0.05; Differences in Least Squares means = -1.9484, 95% CI 2-sided [-4.1009 to 0.2040] — The difference is calculated as Aflibercept minus Ranibizumab. A positive value favors Aflibercept 2mg Q4
Statistical Analysis 2: Comparison: Ranibizumab 0.5mg Q4 vs Aflibercept Injection (EYLEA, VEGF Trap-Eye) 0.5mg Q4; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.9555, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Differences in Least Squares means = -0.0620, 95% CI 2-sided [-2.2398 to 2.1158] — The difference is calculated as Aflibercept minus Ranibizumab. A positive value favors Aflibercept 0.5mg Q4
Statistical Analysis 3: Comparison: Ranibizumab 0.5mg Q4 vs Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg Q8; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.4131, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Differences in Least Squares means = -0.9014, 95% CI 2-sided [-3.0615 to 1.2587] — The difference is calculated as Aflibercept minus Ranibizumab. A positive value favors the Aflibercept 2mg Q8 group

3. Secondary Outcome: Percentage of Participants Who Gained at Least 15 Letters of Vision in the ETDRS Letter Score in the Study Eye at Week 52 - LOCF
Description: Defined study baseline range of ETDRS Best Corrected Visual Acuity letter score of 73 to 25 (= Acuity of 20/40 to 20/320) in the study eye; a higher score represents better functioning.
  Nominator = (Number of participants who maintained vision * 100); Denominator = Number of participants analyzed.
Time Frame: At week 52
Population: Full-Analysis Set; imputation technique: LOCF
Measure: Number; unit: Percentage of participants
Arm/Group | Ranibizumab 0.5mg Q4 | Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg Q4 | Aflibercept Injection (EYLEA, VEGF Trap-Eye) 0.5mg Q4 | Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg Q8
Number analyzed (Participants) | 291 | 309 | 296 | 306
Percentage of participants | 34.02 | 29.45 | 34.80 | 31.37
Statistical Analysis 1: Comparison: Ranibizumab 0.5mg Q4 vs Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg Q4; The null hypothesis is that the two proportions are equal; Test type: Superiority or Other; p = 0.229, Chi-squared — [p-value comment as in outcome 2, analysis 1]; Risk Difference (RD) = -4.57, 95% CI 2-sided [-12.02 to 2.88] — The difference is calculated as Aflibercept minus Ranibizumab. A positive value favors the Aflibercept 2mg Q4 group
Statistical Analysis 2: Comparison: Ranibizumab 0.5mg Q4 vs Aflibercept Injection (EYLEA, VEGF Trap-Eye) 0.5mg Q4; The null hypothesis is that the two proportions are equal; Test type: Superiority or Other; p = 0.843, Chi-squared — [p-value comment as in outcome 2, analysis 1]; Risk Difference (RD) = 0.78, 95% CI 2-sided [-6.91 to 8.46] — The difference is calculated as Aflibercept minus Ranibizumab. A positive value favors the Aflibercept 0.5mg Q4 group
Statistical Analysis 3: Comparison: Ranibizumab 0.5mg Q4 vs Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg Q8; The null hypothesis is that the two proportions are equal; Test type: Superiority or Other; p = 0.490, Chi-squared — [p-value comment as in outcome 2, analysis 1]; Risk Difference (RD) = -2.65, 95% CI 2-sided [-10.18 to 4.88] — The difference is calculated as Aflibercept minus Ranibizumab. A positive value favors the Aflibercept 2mg Q8 group

4. Secondary Outcome: Mean Change From Baseline in National Eye Institute 25-item Visual Function Questionnaire (NEI VFQ-25) Total Score at Week 52 - LOCF
Description: The possible range of the NEI VFQ-25 total score is between 0 (worst possible) and 100 (best possible).
Time Frame: Baseline and at week 52
Population: Full-Analysis Set with assessment for this outcome measure; imputation technique: LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ranibizumab 0.5mg Q4 | Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg Q4 | Aflibercept Injection (EYLEA, VEGF Trap-Eye) 0.5mg Q4 | Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg Q8
Number analyzed (Participants) | 287 | 304 | 290 | 299
Scores on a scale | 6.3 (14.8) | 4.5 (15.0) | 5.1 (13.7) | 4.9 (14.7)
Statistical Analysis 1: Comparison: Ranibizumab 0.5mg Q4 vs Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg Q4; The pairwise comparison is performed as contrast statement in the analysis of covariance model with treatment group as fixed factor (all 4 treatment groups) and the baseline NEI VFQ-25 total score as covariate. The null hypothesis is that both mean changes are equal; Test type: Superiority or Other; p = 0.0097, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Differences in Least Squares means = -2.7885, 95% CI 2-sided [-4.9012 to -0.6757] — The difference is calculated as Aflibercept minus Ranibizumab. A positive value favors Aflibercept 2mg Q4
Statistical Analysis 2: Comparison: Ranibizumab 0.5mg Q4 vs Aflibercept Injection (EYLEA, VEGF Trap-Eye) 0.5mg Q4; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.3917, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Differences in Least Squares means = -0.9320, 95% CI 2-sided [-3.0658 to 1.2019] — The difference is calculated as Aflibercept minus Ranibizumab. A positive value favors Aflibercept 0.5mg Q4
Statistical Analysis 3: Comparison: Ranibizumab 0.5mg Q4 vs Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg Q8; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0717, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Differences in Least Squares means = -1.9470, 95% CI 2-sided [-4.0659 to 0.1718] — The difference is calculated as Aflibercept minus Ranibizumab. A positive value favors Aflibercept 2mg Q8

5. Secondary Outcome: Mean Change From Baseline in Choroidal Neovascularization (CNV) Area at Week 52 - LOCF
Description: CNV area values measured in square millimeters; lower values represent better outcomes.
Time Frame: Baseline and at week 52
Population: Full-Analysis Set with assessment for this outcome measure; imputation technique: LOCF
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Ranibizumab 0.5mg Q4 | Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg Q4 | Aflibercept Injection (EYLEA, VEGF Trap-Eye) 0.5mg Q4 | Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg Q8
Number analyzed (Participants) | 278 | 294 | 287 | 289
mm^2 | -4.16 (5.90) | -5.95 (6.12) | -4.24 (6.13) | -5.16 (5.87)
Statistical Analysis 1: Comparison: Ranibizumab 0.5mg Q4 vs Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg Q4; The pairwise comparison is performed as contrast statement in the analysis of covariance model with treatment group as fixed factor (all 4 treatment groups) and the baseline CNV area as covariate. The null hypothesis is that both mean changes are equal; Test type: Superiority or Other; p = 0.0038, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Differences in Least Squares means = -1.180, 95% CI 2-sided [-1.979 to -0.382] — The difference is calculated as Aflibercept minus Ranibizumab. A negative value favors Aflibercept 2mg Q4
Statistical Analysis 2: Comparison: Ranibizumab 0.5mg Q4 vs Aflibercept Injection (EYLEA, VEGF Trap-Eye) 0.5mg Q4; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.6784, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Differences in Least Squares means = 0.170, 95% CI 2-sided [-0.632 to 0.972] — The difference is calculated as Aflibercept minus Ranibizumab. A negative value favors Aflibercept 0.5mg Q4
Statistical Analysis 3: Comparison: Ranibizumab 0.5mg Q4 vs Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg Q8; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0727, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Differences in Least Squares means = -0.733, 95% CI 2-sided [-1.534 to 0.068] — The difference is calculated as Aflibercept minus Ranibizumab. A negative value favors Aflibercept 2mg Q8

ADVERSE EVENTS:
Arm/Group | Ranibizumab 0.5mg Q4 | Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg Q4 | Aflibercept Injection (EYLEA, VEGF Trap-Eye) 0.5mg Q4 | Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg Q8
Serious Adverse Events (participants affected / at risk) | 65/291 | 81/309 | 72/297 | 81/307
Other Adverse Events (participants affected / at risk) | 254/291 | 259/309 | 251/297 | 260/307
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab 0.5mg Q4 (N=291) | Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg Q4 (N=309) | Aflibercept Injection (EYLEA, VEGF Trap-Eye) 0.5mg Q4 (N=297) | Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg Q8 (N=307)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 2
Angina pectoris (Cardiac disorders) | 1 | 1 | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 1 | 0
Aortic valve stenosis (Cardiac disorders) | 1 | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 2 | 2 | 3
Atrial flutter (Cardiac disorders) | 0 | 2 | 1 | 1
Atrioventricular block (Cardiac disorders) | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0 | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 1 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0
Coronary artery thrombosis (Cardiac disorders) | 1 | 0 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 4 | 3 | 3 | 4
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 2
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 2 | 2 | 2
Cardiac disorder (Cardiac disorders) | 0 | 0 | 1 | 0
Mitral valve disease (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiovascular insufficiency (Cardiac disorders) | 0 | 0 | 0 | 2
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Tympanic membrane disorder (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Blindness (Eye disorders) | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 5 | 4 | 4 | 4
Cataract cortical (Eye disorders) | 1 | 0 | 0 | 0
Cataract nuclear (Eye disorders) | 0 | 1 | 1 | 0
Cataract subcapsular (Eye disorders) | 0 | 1 | 0 | 0
Choroidal detachment (Eye disorders) | 0 | 0 | 0 | 1
Hyphaema (Eye disorders) | 1 | 0 | 0 | 0
Iridocyclitis (Eye disorders) | 0 | 0 | 0 | 1
Macular cyst (Eye disorders) | 0 | 0 | 0 | 1
Macular degeneration (Eye disorders) | 0 | 1 | 0 | 3
Maculopathy (Eye disorders) | 0 | 0 | 0 | 1
Posterior capsule opacification (Eye disorders) | 2 | 0 | 0 | 0
Retinal degeneration (Eye disorders) | 1 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 3 | 0 | 1 | 0
Retinal haemorrhage (Eye disorders) | 4 | 3 | 4 | 2
Retinal pigment epitheliopathy (Eye disorders) | 0 | 1 | 0 | 0
Retinal vein occlusion (Eye disorders) | 0 | 1 | 0 | 0
Visual acuity reduced (Eye disorders) | 3 | 5 | 1 | 7
Vitreous detachment (Eye disorders) | 0 | 0 | 0 | 1
Vitreous haemorrhage (Eye disorders) | 1 | 1 | 0 | 0
Macular hole (Eye disorders) | 0 | 0 | 1 | 0
Ocular retrobulbar haemorrhage (Eye disorders) | 0 | 0 | 0 | 1
Choroidal neovascularisation (Eye disorders) | 1 | 1 | 0 | 2
Retinal pigment epithelial tear (Eye disorders) | 1 | 0 | 1 | 2
Macular scar (Eye disorders) | 0 | 1 | 0 | 0
Age-related macular degeneration (Eye disorders) | 0 | 3 | 0 | 1
Abdominal mass (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abnormal faeces (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Colonic polyp (Gastrointestinal disorders) | 2 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Femoral hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Femoral hernia, obstructive (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Rectal polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Rectal prolapse (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Enterovesical fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Bowel movement irregularity (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 1
Chest pain (General disorders) | 3 | 1 | 1 | 1
Chills (General disorders) | 0 | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 1 | 0
Hernia (General disorders) | 0 | 0 | 1 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0
Multi-organ failure (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 2 | 0 | 1
Disease progression (General disorders) | 0 | 1 | 0 | 0
Device malfunction (General disorders) | 0 | 1 | 0 | 0
Device dislocation (General disorders) | 1 | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 2 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 2 | 2 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 1 | 1
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0
Endophthalmitis (Infections and infestations) | 0 | 1 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 1
Gastroenteritis salmonella (Infections and infestations) | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 1
Herpes zoster ophthalmic (Infections and infestations) | 0 | 0 | 0 | 1
Liver abscess (Infections and infestations) | 0 | 1 | 0 | 0
Peridiverticular abscess (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 4 | 2 | 6
Pneumonia pneumococcal (Infections and infestations) | 0 | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 2 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 0
Dysentery (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis norovirus (Infections and infestations) | 1 | 0 | 0 | 0
Accident (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Burns second degree (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Cerebral haemorrhage traumatic (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 3
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1
Skull fractured base (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Graft thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Traumatic brain injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 2 | 1 | 3 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Spinal column injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Blood osmolarity decreased (Investigations) | 0 | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0 | 0
Haematocrit decreased (Investigations) | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 0
Intraocular pressure increased (Investigations) | 0 | 0 | 1 | 2
Mean cell haemoglobin decreased (Investigations) | 0 | 1 | 0 | 0
Mean cell volume decreased (Investigations) | 0 | 1 | 0 | 0
Red blood cell count decreased (Investigations) | 0 | 1 | 0 | 0
Investigation (Investigations) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | 0
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Bladder cancer stage 0, with cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 3 | 1
Carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Colon cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Metastases to ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 2 | 1 | 2
Dementia Alzheimer's type (Nervous system disorders) | 0 | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 1
Hypertensive encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Normal pressure hydrocephalus (Nervous system disorders) | 0 | 1 | 0 | 0
Petit mal epilepsy (Nervous system disorders) | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 1 | 0 | 1
Syncope (Nervous system disorders) | 1 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 2 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 1 | 0 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 1 | 0 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Lacunar infarction (Nervous system disorders) | 0 | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 1
Nerve root compression (Nervous system disorders) | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 3 | 0 | 2
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1
Cystitis noninfective (Renal and urinary disorders) | 0 | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pemphigus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Blepharoplasty (Surgical and medical procedures) | 0 | 1 | 0 | 0
Strangulated hernia repair (Surgical and medical procedures) | 0 | 0 | 1 | 0
Surgery (Surgical and medical procedures) | 0 | 1 | 0 | 0
Hip surgery (Surgical and medical procedures) | 0 | 0 | 0 | 1
Haematoma evacuation (Surgical and medical procedures) | 1 | 0 | 0 | 0
Vaginal operation (Surgical and medical procedures) | 1 | 0 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 1 | 1 | 1
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 1
Hypertensive crisis (Vascular disorders) | 1 | 1 | 0 | 2
Varicose vein (Vascular disorders) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Peripheral artery aneurysm (Vascular disorders) | 0 | 0 | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab 0.5mg Q4 (N=291) | Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg Q4 (N=309) | Aflibercept Injection (EYLEA, VEGF Trap-Eye) 0.5mg Q4 (N=297) | Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg Q8 (N=307)
Atrioventricular block first degree (Cardiac disorders) | 16 | 25 | 23 | 22
Cataract (Eye disorders) | 29 | 36 | 34 | 32
Conjunctival haemorrhage (Eye disorders) | 34 | 33 | 46 | 35
Conjunctivitis (Eye disorders) | 19 | 14 | 8 | 21
Dry eye (Eye disorders) | 14 | 12 | 15 | 16
Eye pain (Eye disorders) | 28 | 36 | 25 | 24
Macular cyst (Eye disorders) | 18 | 8 | 9 | 9
Macular degeneration (Eye disorders) | 37 | 35 | 42 | 51
Macular oedema (Eye disorders) | 17 | 16 | 23 | 22
Maculopathy (Eye disorders) | 13 | 16 | 18 | 10
Ocular hyperaemia (Eye disorders) | 20 | 18 | 17 | 10
Retinal cyst (Eye disorders) | 13 | 20 | 17 | 13
Retinal degeneration (Eye disorders) | 33 | 37 | 27 | 23
Retinal haemorrhage (Eye disorders) | 82 | 84 | 70 | 82
Retinal oedema (Eye disorders) | 34 | 32 | 31 | 40
Retinal pigment epitheliopathy (Eye disorders) | 28 | 23 | 20 | 28
Visual acuity reduced (Eye disorders) | 46 | 44 | 55 | 60
Vitreous detachment (Eye disorders) | 22 | 30 | 17 | 24
Conjunctival hyperaemia (Eye disorders) | 18 | 8 | 11 | 5
Detachment of retinal pigment epithelium (Eye disorders) | 38 | 37 | 33 | 31
Choroidal neovascularisation (Eye disorders) | 28 | 25 | 28 | 23
Age-related macular degeneration (Eye disorders) | 26 | 28 | 26 | 38
Diarrhoea (Gastrointestinal disorders) | 14 | 9 | 16 | 16
Pyrexia (General disorders) | 19 | 12 | 19 | 8
Bronchitis (Infections and infestations) | 13 | 17 | 20 | 12
Influenza (Infections and infestations) | 14 | 19 | 12 | 23
Nasopharyngitis (Infections and infestations) | 39 | 25 | 32 | 26
Blood glucose increased (Investigations) | 9 | 17 | 14 | 18
Intraocular pressure increased (Investigations) | 37 | 38 | 24 | 29
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 8 | 15 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 17 | 19 | 12 | 16
Dizziness (Nervous system disorders) | 15 | 8 | 4 | 5
Headache (Nervous system disorders) | 14 | 12 | 16 | 20
Hypertension (Vascular disorders) | 42 | 41 | 33 | 34

LIMITATIONS AND CAVEATS:
The conditional sequence of hypothesis testing had to stop after testing the first superiority hypothesis. Therefore, all further statistical tests are exploratory tests.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Confidentiality agreement with sponsor, contract with the sponsor via the CRO (Clinical research organization), set up based on local legal requirements, changes addressed+confirmed with local responsible persons; PIs interested in presenting the study on meetings, contacted the sponsor and received slides and approval to do so either by the Clinical Lead or the Medical Affairs department